CLINICAL TRIAL: NCT06597825
Title: Antibacterial Effect of Sodium Hypochlorite Combined With Etidronic Acid in Apical Periodontitis Treatment: A Prospective, Single Blinded, Randomised Clinical Trial
Brief Title: Antibacterial Effect of NaOCl With Etidronic Acid in Apical Periodontitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Pelin Tufenkci, Associate Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clinical Research-2019/37
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Bacterial reduction; etidronic acid; root canal irrigation; sodium hypochlorite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- İrrigation protocols (Group I) (Experimental): Group I: the root canal was irrigated with 1 ml of 17% EDTA (Microvem, Istanbul, Turkey), and the solution was kept in the canal for 1 minute. The canal was subsequently irrigated with 2 ml of distilled water and 3 ml of 2.5% NaOCl for 1 minute.
  Interventions: Drug: root canal irrigation solutions (NaOCl+EDTA, NaOCl+HEDP)
- İrrigation protocols (Group II) (Experimental): Group II: HEDP (DualRinse HEDP, Medcem, Vienna, Austria), containing 0.9 mg of etidronic acid per capsule, was added to 10 ml of 2.5% NaOCl in a sterile container according to the manufacturer's instructions. The solution, which was prepared just before use in the canal, was mixed for 1 min to ensure that the powder was fully dissolved. The canal was then irrigated with 4 ml of the 2.5% NaOCl - 9% HEDP combined solution for 2 minutes.
  Interventions: Drug: root canal irrigation solutions (NaOCl+EDTA, NaOCl+HEDP)
- İrrigation protocols (Group III) (Experimental): Group III: A similar irrigation protocol to that of Group I was followed, with an additional 1-minute sonic activation using the EA device on 3 ml of 2.5% NaOCl. The tip of the EA was placed 2 mm away from the WL and the irrigant was activated with 10,000 cycles per minute with a tip size 0.04/35.
  Interventions: Drug: root canal irrigation solutions (NaOCl+EDTA, NaOCl+HEDP)
- İrrigation protocols (Group IV) (Experimental): Group IV: Similar to Group II, the canal was filled with 4 ml of the 2.5% NaOCl - 9% HEDP combined solution for 1 minute. The tip of the EA was placed 2 mm away from the WL, followed by 1 minute of sonic activation with the EA device (10,000 cycles per minute with a tip size 0.04/35).
  Interventions: Drug: root canal irrigation solutions (NaOCl+EDTA, NaOCl+HEDP)

INTERVENTIONS:
Drug: root canal irrigation solutions (NaOCl+EDTA, NaOCl+HEDP) — After cavity preparation with sterile burs, rubber dam components were applied to the tooth. The root canal filling material was removed via retreatment files. After the working length was determined, in all the groups, the canals were filled with distilled water. S1were taken from the canal after retreatment. Irrigation protocols were applied for 4 groups. S2 were taken from the canal. Intracanal medicament was placed in the root canal, the cavity was securely sealed. After 14 days,the medicament was removed with 10 mL of 17% EDTA and subsequently irrigated with 5 ml of distilled water, S3 was taken by sterile paper points. The final irrigation was performed according to the group to which the tooth belonged, and S4 was collected as before. the root canals were dried with sterile paper points and filled gutta-percha master cones and sealer.
  Other Names: Root canal irrigation activation (Endoactivator) (Device)

SUMMARY:
Sodium hypochlorite (NaOCl), the most commonly used irrigation solution during chemomechanical preparation, plays a significant role in eliminating bacteria within root canals. Additionally, after preparation with different concentrations of NaOCl, 30% to 70% resistant bacteria were observed in the root canals. For this reason, new protocols have been developed to increase the effectiveness of NaOCl in chemomechanical preparation and to support disinfection within root canals. Recently, etidronic acid (1-hydroxyethane 1,1-diphosphonic acid [HEDP]), a biocompatible chelating agent, has emerged as an alternative irrigation solution. It has been suggested to combine and use this solution with NaOCl.

This study aims to evaluate the antimicrobial effectiveness of NaOCl in the root canal, which is used in combination with HEDP or sequentially with Ethylenediaminetetraacetic acid (EDTA) in the final irrigation after retreatment. Additionally, the effect of activation with Endoactivator (EA) on microbial reduction was assessed.

ELIGIBILITY:
Inclusion Criteria:

The study included teeth from patients aged 18-65 years who had no systemic disease and had not undergone antibiotic therapy in the past three months. To ensure standardization, all the treatments were performed by a single clinician.

1. A minimum of 2 years since the initial root canal treatment
2. Single rooted mandibular premolar with apical periodontitis (AP) and a canal filling within 4 mm from the apex on radiographic examination
3. The absence of pain on palpation and percussion, healthy periodontal tissues, and no mobility,
4. Presence of a coronal restoration (teeth that have not retained permanent restoration over the previous root canal treatment).

Exclusion Criteria:

1. Patients who have received antibiotic therapy in the last 3 months,
2. Patients with diabetes, pregnancy, immunosuppression and cardiovascular disease,
3. Absence of a coronal restoration
4. Presence of pain on palpation and percussion, mobility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Total bacterial load (CFU/ml) in root canal samples of teeth | From enrollment to the end of treatment at 2 weeks
  In all the groups, A sterile paper point of size R50 was placed at the working length (WL) and left in the canal for 1 minute. Three paper points were then placed into an Eppendorf tube containing phosphate-buffered saline (PBS). The samples taken from the canal after retreatment were recorded as the S1. After root canal preparation and irrigation protocols, S2 sample was taken. After dried protocol, medicament was placed in the root canal.After 14 days,the intracanal medicament was removed with 17% EDTA. The root canal was irrigated with 5 ml of distilled water.S3 was taken by sterile R50 paper points. The final irrigation was performed according to the group to which the tooth belonged,the S4 was collected as before.Each sample obtained from the patient was placed into culture medium.The inoculated plates were incubated at 37°C for 48 hours. After incubation, the total bacterial counts were determined by calculating the number of colony-forming units (CFU/ml) on the plates.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University Dentistry Faculty Department of Endodontics, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Siqueira JF Jr, Rôças IN. Clinical implications and microbiology of bacterial persistence after treatment procedures. J Endod 2008;34:1291-12301.e3. 2. Ricucci D, Siqueira JF Jr, Bate AL, Pitt Ford TR. Histologic investigation of root canal-treated teeth with apical periodontitis: a retrospective study from twenty-four patients. J Endod 2009;35:493-502. 3. Zandi H, Petronijevic N, Mdala I, et al. Outcome of endodontic retreatment using 2 root canal irrigants and influence of infection on healing as determined by a molecular method: a randomized clinical trial. J Endod 2019;45:1089-10898.e5. 4. Rodrigues RCV, Zandi H, Kristoffersen AK, Enersen M, Mdala I, Ørstavik D, Rôças IN, Siqueira JF Jr. Influence of the Apical Preparation Size and the Irrigant Type on Bacterial Reduction in Root Canal-treated Teeth with Apical Periodontitis. J Endod. 2017 Jul;43(7):1058-1063. 5. Rôças IN, Provenzano JC, Neves MA, Siqueira JF Jr. Disinfecting Effects of Rotary Instrumentation with Either 2.5% Sodium Hypochlorite or 2% Chlorhexidine as the Main Irrigant: A Randomized Clinical Study. J Endod. 2016 Jun;42(6):943-7. 6. Paiva SS, Siqueira JF Jr, Rôças IN, Carmo FL, Ferreira DC, Curvelo JA, Soares RM, Rosado AS. Supplementing the antimicrobial effects of chemomechanical debridement with either passive ultrasonic irrigation or a final rinse with chlorhexidine: a clinical study. J Endod. 2012 Sep;38(9):1202-6. 7. Siqueira JF Jr, Rôças IN. Optimizing single-visit disinfection with supplementary approaches: a quest for predictability. Aust Endod J 2011;37:92-8.